CLINICAL TRIAL: NCT02760251
Title: Thrombopoietin-receptor Agonist-immunomodulation in Young Adult Primary Immune Thrombocytopenia (ITP): A Multi-center Open Label Trial With Romiplostim
Brief Title: Immunomodulation With Romiplostim in Young Adults With ITP
Acronym: iROM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20149180
Record Dates: First submitted 2016-04-15; First posted 2016-05-03 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Immune Thrombocytopenia
Keywords: immunomodulation
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Romiplostim (a thrombopoietin-receptor agonist, TPO-RA) will be administered subcutaneously once weekly over 22 weeks with a starting dose of 1mcg/kg body weight. The dose will be adjusted based on platelet counts as described in the summary of Product Characteristics (SmPC). Followup examination at week 52.
  Interventions: Drug: romiplostim

INTERVENTIONS:
Drug: romiplostim
  Other Names: Nplate

SUMMARY:
The study aims to investigate immunomodulatory effects of thrombopoietin-receptor Agonist (TPO-RA) in patients with primary ITP, who failed first-line therapy or who became intolerant to it. It is hypothesized that the early phase of this autoimmune disease may exhibit a stronger immunomodulatory potential in response to a stimulus, such as romiplostim. Such a process may subsequently be capable to induce regulatory mechanisms or tolerance.

Romiplostim (a thrombopoietin-receptor agonist, TPO-RA) will be administered subcutaneously once weekly over 22 weeks with a starting dose of 1mcg/kg body weight. The dose will be adjusted based on platelet counts as described in the summary of Product Characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (see informed consent form)
* Primary ITP according to the definition of Rodeghiero et al. (52) and a platelet count of <30x109/l
* Age range: 18-45 years
* Previously treated patients, with failure or intolerance to first-line therapy, or relapse after first-line therapy, i.e. corticosteroids, intravenous immunoglobulin (IVIG), or anti-D immunoglobulins

Exclusion Criteria:

* Adults older than 45 and children younger than 18 years
* Platelet count higher than 30x109/l at time of screening
* Suspicion of secondary ITP
* Positive family history for ITP
* Presence or history of autoimmune disease as judged by the investigator
* Hepatosplenomegaly
* Presence or history of relevant hepatic disease as judged by the investigator
* Presence or history of thromboembolic disease as judged by the investigator
* Patients with splenectomy
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe double contraception (see 7.1)
* Any vaccination 2 weeks prior start of the study
* Drugs with a known impact on the immune system or on platelet function must be recorded and an exclusion of the study should be discussed with the study center
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia of the study subject
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Previous treatment with romiplostim or eltrombopag
* Hypersensitivity to the active substance or to any of the excipients or to E. coli derived proteins
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04; Primary Completion 2019-07 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in Interleukin (IL)-4 concentrations (pg/ml) from baseline to week 22 | baseline and 22 weeks
  The primary aim of the study is to demonstrate an immunomodulatory effect of the study drug. Investigators expect a shift in the Th1/Th2 balance towards Th2.
  The primary outcome is to compare the pre- and post-treatment IL-4 concentrations (pg/ml) of all included patients (Th2 profile). Assessment of change in pre- and post-treatment IL-4 concentrations (pg/ml).

SECONDARY OUTCOMES:
Change in immunomodulation as assessed by immune cell characteristics between baseline and week 22 | baseline and 22 weeks
  Immunologic parameters will be investigated between baseline and week 22 of the study: immune cell characteristics
  fluorescence-activated cell sorting (FACS): B cells: cluster of Differentiation Antigen (CD)3- cluster of Differentiation Antigen (CD)19+ Memory B lymphocytes CD19+cluster of Differentiation Antigen (CD)10-cluster of Differentiation Antigen (CD)27+cluster of Differentiation Antigen (CD)38- Plasma cells: CD19+ CD10- cluster of Differentiation Antigen (CD)20- CD27++ cluster of Differentiation Antigen (CD)38++ Tcells and subpopulations: CD3+/ CD3+ CD4+/ CD3+ cluster of Differentiation Antigen (CD)8+ natural killer (NK) cells CD3- cluster of Differentiation Antigen (CD)16+ cluster of Differentiation (CD)56+ Monocytes CD56- cluster of Differentiation Antigen (CD)14 (low) CD16+ cluster of Differentiation Antigen (CD)33 Tregs CD4+ cluster of Differentiation Antigen (CD)25 superhigh FoxP3+
Change in immunomodulation as assessed by immune cell characteristics between baseline and week 10 | baseline and 10 weeks
  Immunologic parameters will be investigated between baseline and week 10 of the study: immune cell characteristics
  FACS:
  B cells: CD3- CD19+ Memory B lymphocytes CD19+CD10-CD27+CD38- Plasma cells: CD19+ CD10- CD20- CD27++ CD38++ Tcells and subpopulations: CD3+/ CD3+ CD4+/ CD3+ CD8+ NK cells CD3- CD16+ CD56+ Monocytes CD56- CD14 (low) CD16+ CD33 Tregs CD4+ CD25 superhigh FoxP3+
Change in immunomodulation as assessed by messenger ribonucleic acid (mRNA) of cytokines between baseline and week 22 | baseline and 22 weeks
  mRNA of cytokines will be investigated between baseline and week 22
  mRNA essays (real-time quantitative PCR): cytokine mRNA (interleucin (IL)2, interleucin (IL)4, interleucin (IL)6, interleucin (IL)10, IL17, interleucin (IL)35, IFNgamma, TNFalpha, transforming growth factor (TGF)-β)
Change in immunomodulation as assessed by mRNA of immune cells between baseline and week 22 | baseline and 22 weeks
  mRNA of immune cells will be investigated between baseline and week 22
  mRNA essays (real-time quantitative PCR): mRNA Th1 (T-bet), Th2 (GATA-3), Th17 (RORγt), Tregs (Foxp3)
Change in immunomodulation as assessed by mRNA of cytokines between baseline and week 10 | baseline and 10 weeks
  mRNA of cytokines will be investigated between baseline and week 10
  mRNA essays (real-time quantitative PCR): cytokine mRNA (IL2, IL4, IL6, IL10, IL17, IL35, IFNgamma, TNFalpha, TGF-β)
Change in immunomodulation as assessed by mRNA of immune cells between baseline and week 10 | baseline and 10 weeks
  mRNA of immune cells will be investigated between baseline and week 10
  mRNA essays (real-time quantitative PCR): mRNA Th1 (T-bet), Th2 (GATA-3), Th17 (RORγt), Tregs (Foxp3)
Change in immunomodulation as assessed by cytokine concentrations between baseline and week 22 | baseline and 22 weeks
  cytokine concentration will be investigated between baseline and week 22
  ELISA Cytokines: IL2, IL4, IL6, IL10, IL17, IL35, IFNgamma, TNFalpha, TGF- β
Change in immunomodulation as assessed by cytokine concentrations between baseline and week 10 | baseline and 10 weeks
  cytokine concentration will be investigated between baseline and week 10
  ELISA Cytokines: IL2, IL4, IL6, IL10, IL17, IL35, IFNgamma, TNFalpha, TGF- β
Clinical response between baseline and week 52: number of severe bleeding | baseline and 52 weeks
  Clinical characterization of response to romiplostim therapy will be assessed additionally : measurement of severe bleeding (score Bolton-Maggs)
Clinical response between baseline and week 52: number of days in hospital | baseline and 52 weeks
  Clinical characterization of response to romiplostim therapy will be assessed additionally : need of inpatient daycare
Clinical response between baseline and week 52: platelet more than >100G/l | baseline and 52 weeks
  Clinical characterization of response to romiplostim therapy will be assessed additionally : assessment of platelet response to romiplostim, according to the definitions of Rodeghiero et al. (49).
Change in immunomodulation as assessed by immune cell characteristics between baseline and week 52 | baseline and 52 weeks
  Immunologic parameters will be investigated between baseline and week 52 of the study: immune cell characteristics
  FACS:
  B cells: CD3- CD19+ Memory B lymphocytes CD19+CD10-CD27+CD38- Plasma cells: CD19+ CD10- CD20- CD27++ CD38++ Tcells and subpopulations: CD3+/ CD3+ CD4+/ CD3+ CD8+ NK cells CD3- CD16+ CD56+ Monocytes CD56- CD14 (low) CD16+ CD33 Tregs CD4+ CD25 superhigh FoxP3+
Change in immunomodulation as assessed by mRNA of immune cells between baseline and week 52 | baseline and 52 weeks
  mRNA of immune cells will be investigated between baseline and week 52
  mRNA essays (real-time quantitative PCR): mRNA Th1 (T-bet), Th2 (GATA-3), Th17 (RORγt), Tregs (Foxp3)
Change of immunomodulation as assessed by mRNA of cytokines between baseline and week 52 | baseline and 52 weeks
  mRNA of cytokines will be investigated between baseline and week 52
  mRNA essays (real-time quantitative PCR): cytokine mRNA (IL2, IL4, IL6, IL10, IL17, IL35, IFNgamma, TNFalpha, TGF-β)
Change in immunomodulation as assessed by cytokine concentrations between baseline and week 52 | baseline and 52 weeks
  cytokine concentration will be investigated between baseline and week 52
  ELISA Cytokines: IL2, IL4, IL6, IL10, IL17, IL35, IFNgamma, TNFalpha, TGF- β
Clinical response between baseline and week 52: frequency of use of rescue treatment | baseline and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kühne, Prof.Dr.med, Principal Investigator — UKBB
Locations (5):
- Switzerland (5):
  - Liestal Cantonal Hospital, Liestal, Basel-Landschaft
  - Lucerne Cantonal Hospital, Lucerne, Canton of Lucerne
  - Aarau Cantonal Hospital, Aarau
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schifferli A, Rufer A, Rovo A, Nimmerjahn F, Cantoni N, Holbro A, Favre G, Dirks J, Wieland A, Faeth H, Pereira R, Kuhne T. Immunomodulation with romiplostim as a second-line strategy in primary immune thrombocytopenia: The iROM study. Br J Haematol. 2023 Oct;203(1):119-130. doi: 10.1111/bjh.19074. PMID 37735543